CLINICAL TRIAL: NCT02280122
Title: Activated Matrix Metalloproteinase 8 (aMMP-8) in Saliva as Diagnostic Test for Periodontal Disease? A Case-control Study
Brief Title: Activated MMP-8 as Diagnostic Test for Periodontitis
Acronym: MMP-8
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Peter Eickholz, Prof. Dr. med. dent., Goethe University
Other Study IDs: 144/13
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Generalized Chronic Periodontitis
Keywords: activated matrix metalloproteinase 8; untreated moderate/severe chronic periodontitis; saliva; sensitivity/specificity
MeSH Terms: conditions — Chronic Periodontitis; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- gen. mod. to sev. chronic periodontitis: * Sites with probing pocket depths (PPD) ≥ 3.5 mm
  * Attachment loss (PAL-V) ≥ 3 mm > 30% of sites
  * no Intervention provided
- periodontally healthy: * PPD ≤ 3 mm
  * PAL-V ≤ 2 mm at < 30% of sites
  * BOP < 20%
  * No radiographically detectable bone loss: distance cemento-enamel junction to provided
  * no Intervention but aMMP-8 test
  Interventions: Other: no intervention provided

INTERVENTIONS:
Other: no intervention provided — No Intervention was rendered but the aMMP-8 test was made
  Groups: periodontally healthy

SUMMARY:
Background: Untreated periodontal disease may influence general health. However, how may a physician who is not trained in periodontal probing detect untreated periodontitis? Activated matrix metalloproteinase-8 (aMMP-8) in saliva correlates with periodontal probing parameters. Thus, sensitivity and specificity of a chair-side test for activated matrix metalloproteinase-8 to detect periodontitis was evaluated.

Methods: Thirty cases (untreated chronic periodontitis; 15 generalized moderate and 15 generalized severe) and 30 controls (probing pocket depths ≤ 3 mm, vertical probing attachment level ≤ 2 mm at < 30% of sites) were examined periodontally. Further, the activated matrix metalloproteinase-8 test was performed. The test kit becomes positive with ≥ 25 ng/ml activated matrix metalloproteinase-8 in the sample.

DETAILED DESCRIPTION:
.The hypotheses behind this study were:

- The aMMP-8 test discriminates between individuals with and without untreated generalized chronic periodontitis

Thus, sensitivity and specificity of a chair-side test for activated matrix metalloproteinase-8 to distinguish between individuals with and without untreated chronic periodontitis as well as between patients with generalized moderate and generalized severe ChP was evaluated.

Patients

A commercially available chair side test to detect increased levels of activated matrix metalloproteinase-8 was used at Dr. Matthias Mayer's dental office (Arndtstr. 14, 60325 Frankfurt am Main) in periodontally healthy individuals and patients with untreated generalized moderate chronic periodontitis (mChP) and generalized severe chronic Periodontitis (sChP).

The companies had provided 70 tests for use. During use the idea arose to retrospectively correlate test results and clinical diagnoses. Thus, a study protocol was submitted to the ethics committee of the Medical Faculty of the Johann Wolfgang Goethe-University Frankfurt/Main. All patients that were examined prior to the vote of the ethics committee were evaluated retrospectively. All following patients were recruited prospectively.

All patients were asked about current smoking (yes/no) and education level (basic school, high school, university). The study complied with the rules of the Declaration of Helsinki and was approved by the Institutional Review Board for Human Studies of the Medical Faculty of the Goethe-University Frankfurt/Main (Application# 144/13).

Chair side test

For all periodontitis patients the activated matrix metalloproteinase-8 test was performed at least 24 hours after clinical examination. For periodontally healthy controls the test was done within a week after clinical examination. First of all patients rinsed with tap water for 30 seconds. Then they spat out the water and waited for 1 min. Now patients rinsed with 5ml of purified water for 30 seconds and spat this sample back into the test cup. Approximately 2 ml of the sampled saliva was now taken up with a syringe. After a filter was put onto the syringe 3 drops of the saliva were pressed through the filter into the ELISA kit. After 5 to 10 min the result was read from the test kit. If both the control and test stripes were visible the respective test was positive (i.e. ≥ 25 ng activated matrix metalloproteinase-8 per ml). All test results were photographed with 2fold magnification.

Statistical analysis

The patient was looked upon as statistical unit. The sensitivity and specificity of the aMMP-8 test was defined as the main outcome variables. All other parameters were control variables.

For all individuals, cigarette pack years were calculated. Group frequencies were expressed for sex, current smoking, education, and activated matrix metalloproteinase-8 (positive/negative). Group means and standard deviations were calculated for age and bleeding on probing. Further, for each individual the following variables were calculated to describe the periodontal status.

Comparisons between groups for dichotomous parameters were made by χ² or Fisher's exact test and for all other parameters by Kruskal-Wallis and Mann-Whitney-U test.

Using backward stepwise logistic regression analysis, factors should be identified that were associated with positive activated matrix metalloproteinase-8 tests.

ELIGIBILITY:
Inclusion Criteria:

* At least18 years of age
* Clinical diagnosis of generalized moderate or generalized severe ChP
* At least 5 teeth present per quadrant
* After application to the ethics committee: written informed consent

Exclusion Criteria:

* Requirement of systemic antibiotics for measures that may cause transitory bacteraemia (e.g. pocket probing)
* Nonsurgical or surgical periodontal treatment within the last 12 months prior to PerioMarker® test
* Systemic or topical subgingival antibiotics within the last 6 months prior to PerioMarker® test
* Anti-inflammatory medication (e.g. non-steroidal anti-inflammatory drugs) during the last 3 months prior to PerioMarker® test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Periodontally healthy individuals and patients with untreated generalized moderate and generalized severe ChP from a German dental Office in Frankfurt/Main
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Eickholz, Dr., Study Chair — Johann Wolfgang Goethe-Universität

REFERENCES:
- [Result] Izadi Borujeni S, Mayer M, Eickholz P. Activated matrix metalloproteinase-8 in saliva as diagnostic test for periodontal disease? A case-control study. Med Microbiol Immunol. 2015 Dec;204(6):665-72. doi: 10.1007/s00430-015-0413-2. Epub 2015 Apr 5. PMID 25841875

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate Chronic Periodontitis: * Sites with probing pocket depths (PPD) ≥ 3.5 mm
  * Attachment loss (PAL-V) 3-4 mm > 30% of sites, PAL-V ≥ 5 mm ≤ 30% of sites
  * no Intervention provided
  no intervention provided: No Intervention was rendered but the aMMP-8 test was made
- Severe Chronic Periodontitis: * Sites with probing PPD ≥ 3.5 mm
  * PAL-V ≥ 5 mm > 30% of sites
  * no Intervention provided
  no intervention provided: No Intervention was rendered but the aMMP-8 test was made
- Periodontally Healthy: * PPD ≤ 3 mm
  * PAL-V ≤ 2 mm at < 30% of sites
  * BOP < 20%
  * No radiographically detectable bone loss: distance cemento-enamel junction to provided
  * no Intervention but aMMP-8 test
  no intervention provided: No Intervention was rendered but the aMMP-8 test was made
Period: Overall Study
Arm/Group | Moderate Chronic Periodontitis | Severe Chronic Periodontitis | Periodontally Healthy
Started | 15 | 15 | 30
Completed | 15 | 15 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Generalised Moderate to Severe Chronic Periodontitis: * Sites with probing pocket depths (PPD) ≥ 3.5 mm
  * Attachment loss (PAL-V) ≥ 3 mm > 30% of sites
  * no Intervention provided
  no intervention provided: No Intervention was rendered but the aMMP-8 test was made
- Total: Total of all reporting groups
Arm/Group | Generalised Moderate to Severe Chronic Periodontitis | Periodontally Healthy | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (10.7) | 28.4 (7.9) | 41.2 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 16 | 10 | 26
Region of Enrollment [Number; unit: participants]
  Germany | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of True Positive/Negative aMMP-8 Tests of All Periodontitis Patients (Sensitivity/Specificity)
Description: First off all patients rinsed with tap water for 30 seconds. Then they spat out the water and waited for 1 min. Now patients rinsed with 5ml of purified water for 30 seconds and spat this sample back into the test cup. Approximately 2 ml of the sampled saliva was now sampled with a syringe. After a filter was put onto the syringe 3 drops of the saliva were pressed through the filter into the ELISA kit. After 5 to 10 min the result was read from the test kit [21]. If both the control and test stripes were visible the respective test was positive (i.e. ≥ 25 ng aMMP 8 per ml). The clinical examiner (SIB) judged the results by simple visual inspection. Already a faint test stripe was judged as positive test. All test results were photographed with 2fold magnification. All images of the test were then evaluated by a second examiner (PE) who was blinded for the clinical diagnoses.
Time Frame: 5 minutes
Measure: Number (95% Confidence Interval); unit: percentage of true cases (sens./spec.)
Groups:
- Sensitivity: Generalised Moderate/Severe Chronic Periodontitis: * Sites with probing pocket depths (PPD) ≥ 3.5 mm
  * Attachment loss (PAL-V) ≥ 3 mm > 30% of sites, PAL-V ≥ 5 mm ≤ 30% of sites
  * no Intervention provided
  no intervention provided: No Intervention was rendered but the aMMP-8 test was made
- Specificity: Periodontally Healthy: * PPD ≤ 3 mm
  * PAL-V ≤ 2 mm at < 30% of sites
  * BOP < 20%
  * No radiographically detectable bone loss: distance cemento-enamel junction to provided
  * no Intervention but aMMP-8 test
  no intervention provided: No Intervention was rendered but the aMMP-8 test was made
Arm/Group | Sensitivity: Generalised Moderate/Severe Chronic Periodontitis | Specificity: Periodontally Healthy
Number analyzed (Participants) | 30 | 30
percentage of true cases (sens./spec.) | 87 [68 to 96] | 60 [41 to 77]

ADVERSE EVENTS:
Groups:
- Generalized Moderate to Severe Chronic Periodontitis: * Sites with probing pocket depths (PPD) ≥ 3.5 mm
  * Attachment loss (PAL-V) 3-4 mm > 30% of sites, PAL-V ≥ 5 mm ≤ 30% of sites
  * no Intervention provided
  no intervention provided: No Intervention was rendered but the aMMP-8 test was made
Arm/Group | Generalized Moderate to Severe Chronic Periodontitis | Periodontally Healthy
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
The aMMP-8 test is sensitive to distinguish untreated periodontally diseased from healthy individuals. However, this study does not provide information how clearly the test may distinguish between gingivitis and untreated chronic periodontitis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No